Official Title: Secondary Versus Tertiary Wound Closure in High Risk Gynecologic Abdominal

**Surgical Incisions** 

IRB-Approved Date: 1/5/21

NCT03861065



Department of Obstetrics and Gynecology

# SECONDARY VERSUS TERTIARY WOUND CLOSURE IN HIGH RISK GYNECOLOGIC ABDOMINAL SURGICAL INCISIONS – CCCWFU 04418

Informed Consent Form to Participate in Research Michael G. Kelly, M.D., Principal Investigator

# **SUMMARY**

You are invited to participate in a research study. The purpose of this research is to study an alternative way to close an abdominal wound. Your wound is at higher risk of developing an infection or separation due to multiple factors that your provider can review with you. The standard approach to your wound would be to leave it partially open and let it heal over a period of 3-6 months ("secondary closure"). In this study, we are studying an alternative way ("tertiary closure") to close your wound sooner. If you agree to participate, we would place a loose suture in your wound during surgery. After surgery, in about 4-7 days, we would close the skin edges/wound by tightening this suture.

Your participation in this research will involve 5 visits and last about 5-6 months. We will monitor the status of your wound and also your quality of life during this time. All research studies involve some risks. A risk to this study that you should be aware of is wound infection and additional wound complications. There is the possibility that you may benefit from participation in this study.

Your participation in this study is voluntary. You do not have to participate in this study if you do not want to. There may be other choices available to you. Some other choices may include having your wound closed in the standard procedure. You will not lose any services, benefits, or rights you would normally have if you choose not to participate.

The remainder of this form contains a more complete description of this study. Please read this description carefully. You can ask any questions if you need help deciding whether to join the study. The person in charge of this study is Michael G. Kelly, M.D. If you have questions, suggestions, or concerns regarding this study or you want to withdraw from the study his/her contact information is:

| If you have any questions, suggestions or | concerns about your rig | ghts as a volunteer in this |
|---|---|---|
| research, contact the Institutional Review | Board at | or the Research Subject |
| Advocate at Wake Forest at | | - |

### INTRODUCTION

You are invited to be in a research study. Research studies are designed to gain scientific knowledge that may help other people in the future. You are being asked to take part in this study because you will have abdominal surgery and have what is considered a high-risk wound. Your participation is voluntary. Please take your time in making your decision as to whether or

Version: 01/21/20 



not you wish to participate. Ask your study doctor or the study staff to explain any words or information contained in this informed consent document that you do not understand. You may also discuss the study with your friends and family.

## WHY IS THIS STUDY BEING DONE?

The purpose of this research study is to determine if closing a surgical wound differently is better than the procedure that is currently used. The wound will be closed with what is considered "tertiary intent." This means, rather than leaving the wound open, the wound will be partially closed after surgery, and then completely closed 4-7 days after surgery. We also want to see how this new wound closure process affects your quality of life.

# HOW MANY PEOPLE WILL TAKE PART IN THE STUDY?

There will be 20 people at one (1) research site that will take part in this study.

# WHAT IS INVOLVED IN THE STUDY?

In this study you will have your surgery as you normally would have it. After the surgery, though, you would have your wound closed differently. In the study procedure, the wound will be partially closed rather than being left open. Sutures in the skin will be placed but not closed. A vacuum assisted closure device will be placed over the wound to help healing. After 4-7 days, the vacuum device will be removed, and your doctor will close the wound.

After the wound is closed we will monitor the wound for complications, healing and infection.

We want to determine how this affects your quality of life, so we would like for you to fill out surveys before surgery; 2, 4 and 6 weeks after surgery; and 3 months after the study (follow-up).

# IF YOU TAKE PART IN THIS STUDY, YOU WILL HAVE THE FOLLOWING TESTS AND PROCEDURES: Tertiary Wound Closure

You will have a tertiary wound closure in this study. The method is described above.

### **Quality of Life Questionnaires**

You will fill out questionnaires or surveys that will tell us how this process if influencing your quality of life.

# HOW LONG WILL I BE IN THE STUDY?

You will be in the study for 12 months. Three of these months are considered follow-up. It is after the formal part of the study, but it allows us to keep track of your health, wound healing and quality of life.

You can stop participating at any time. If you decide to stop participating in the study we encourage you to talk to the investigators or study staff first to learn about any potential health or safety consequences. If you decide to stop participating, we would remove the sutures for the tertiary wound closure and we would close your wound in the standard procedure as described in the summary.

Version: 01/21/20 



# WHAT ARE THE RISKS OF THE STUDY?

Being in this study involves some risk to you. You should discuss the risk of being in this study with the study staff. Risks and side effects related to the tertiary wound closure procedure we are studying include:

- Pain/discomfort,
- Infection
- Time for closure of your abdominal would could be longer with tertiary closure
- You could develop a wound infection with tertiary closure. Symptoms of a wound infection could include skin redness, increase in skin temperature, drainage from your wound or fevers or chills. You might be at higher risk of developing a wound infection with tertiary closure compared to secondary closure. Secondary closure is when your wound is left open to heal on its own over time after surgery
- Because we don't know if closing wounds by the tertiary method is more effective than the standard method of wound closure, there is a chance that your outcome may be better or worse than if you had standard wound closure.

## **Risks of Providing Confidential Information**

In addition, there is a slight risk of a breach of confidentiality. We will do our best to protect your confidential information. There also may be other side effects that we cannot predict. You should tell the research staff about all the medications, vitamins and supplements you take and any medical conditions you have. This may help avoid side effects, interactions and other risks.

Taking part in this research study may involve providing information that you consider confidential or private. Efforts, such as coding research records, keeping research records secure and allowing only authorized people to have access to research records, will be made to keep your information safe.

### Risks of Quality of Life Questionnaires

While filling out quality of life questionnaires, you may experience the feelings or emotions that are being asked about more intensely than you normally would.

# Reproductive Risks and other Issues to Participating in Research

Pregnant women are excluded from participation in this study. If you are a sexually active woman of childbearing potential and have not been using a reliable method of birth control, two negative pregnancy tests performed 15 days apart are required to check for possible early pregnancy prior to starting treatment.

# ARE THERE BENEFITS TO TAKING PART IN THE STUDY?

If you agree to take part in this study, there may or may not be direct benefit to you. We hope the information learned from this study will benefit other people in the future. The benefits of participating in this study may be: a quicker wound closure and improved quality of life.

Version: 01/21/20 Page **3** of **8** 



# WHAT OTHER CHOICES ARE THERE?

You do not have to be in this study to receive treatment. You should talk to your doctor about all the choices you have. Instead of being in this study, you have these options: Wound closure by our standard techniques. The standard for your wound is secondary closure. This means a portion of the wound would be left open to heal on its own over time. This typically takes 3-6 months and requires daily wound care with frequent nursing and doctor's visits.

# WHAT ARE THE COSTS?

Taking part in this study may lead to added costs to you or your insurance company. We will give you an estimate of what the added cost may be based on your particular situation and insurance coverage.

# WILL YOUR RESEARCH RECORDS BE CONFIDENTIAL?

The results of this research study may be presented at scientific or medical meetings or published in scientific journals. Your identity and/or your personal health information will not be disclosed unless it is authorized by you, required by law, or necessary to protect the safety of yourself or others. There is always some risk that even de-identified information might be re-identified.

Participant information may be provided to Federal and other regulatory agencies as required. The Food and Drug Administration (FDA), for example, may inspect research records and learn your identity if this study falls within its jurisdiction.

The purpose of this research study is to obtain data or information on the safety and effectiveness of the tertiary closure technique in abdominal wounds; the results will be provided to the sponsor, the Food and Drug Administration and other federal and regulatory agencies as required.

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. The researchers with this Certificate may not disclose or use information, documents, or biospecimens that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, or be used as evidence, for example, if there is a court subpoena, unless you have consented for this use. Information, documents, or biospecimens protected by this Certificate cannot be disclosed to anyone else who is not connected with the research except, if there is a federal, state, or local law that requires disclosure (such as to report child abuse or communicable diseases but not for federal, state, or local civil, criminal, administrative, legislative, or other proceedings, see below); if you have consented to the disclosure, including for your medical treatment; or if it is used for other scientific research, as allowed by federal regulations protecting research subjects.

The Certificate cannot be used to refuse a request for information from personnel of the United States federal or state government agency sponsoring the project that is needed for auditing or program evaluation by National Institutes of Health, which is funding this project or for information that must be disclosed in order to meet the requirements of the federal Food and Drug Administration (FDA). You should understand that a Certificate of Confidentiality does

Version: 01/21/20 Page **4** of **8** 



not prevent you from voluntarily releasing information about yourself or your involvement in this research. If you want your research information released to an insurer, medical care provider, or any other person not connected with the research, you must provide consent to allow the researchers to release it.

# WILL YOU BE PAID FOR PARTICIPATING?

You will receive no payment or other compensation for taking part in this study. However, you will have parking validation for any study related visits.

The findings from this research may result in the future development of products that are of commercial value. There are no plans to provide you with financial compensation or for you to share in any profits if this should occur.

# WHO IS SPONSORING THIS STUDY?

This study is being sponsored by <u>Wake Forest University Health Sciences</u>. The sponsor is providing money or other support to Wake Forest University Health Sciences to help conduct this study. The researchers do not, however, hold a direct financial interest in the sponsor or the product being studied.

# WHAT HAPPENS IF YOU EXPERIENCE AN INJURY OR ILLNESS AS A RESULT OF PARTICIPATING IN THIS STUDY?

Should you experience a physical injury or illness as a direct result of your participation in this study, Wake Forest University School of Medicine maintains limited research insurance coverage for the usual and customary medical fees for reasonable and necessary treatment of such injuries or illnesses. To the extent research insurance coverage is available under this policy the reasonable costs of these necessary medical services will be paid, up to a maximum of \$25,000. Wake Forest University Baptist Medical Center holds the insurance policy for this coverage. It provides a maximum of \$25,000 coverage for each claim and is limited to a total of \$250,000 for all claims in any one year. The Wake Forest University School of Medicine, and the North Carolina Baptist Hospitals, Incorporated do not assume responsibility to pay for these medical services or to provide any other compensation for such injury or illness. Additional information may be obtained from the Medical Center's Director of Risk and Insurance Management, at

If you are injured, the insurer may require information such as your name, social security number, and date of birth in order to pay for your care. This is because the insurer is required by law to report any payments made to cover the care of any persons who are members of a government insurance plan to the Department of Health and Human Services.

You do not give up any legal rights as a research participant by signing this consent form. For more information on medical treatment for research related injuries or to report a study related illness, adverse event, or injury you should call Michael G. Kelly, M.D. at

# WHAT ABOUT MY HEALTH INFORMATION?

In this research study, any new information we collect from you and/or information we get from your medical records or other facilities about your health or behaviors is considered <u>Protected</u>

Version: 01/21/20 



<u>Health Information</u>. The information we will collect for this research study includes: demographic information, information about your surgery, response to the tertiary closure method, and disease information.

If this research study involves the diagnosis or treatment of a medical condition, then Protected Health Information collected from you during this study will be placed in your medical record, and may be used to help treat you, arrange payment for your care, or assist with Medical Center operations.

We will make every effort to keep your Protected Health Information private. We will store records of your Protected Health Information in a cabinet in a locked office or on a password protected computer.

Your personal health information and information that identifies you ("your health information") may be given to others during and after the study. This is for reasons such as to carry out the study, to determine the results of the study, to make sure the study is being done correctly, to provide required reports and to get approval for new products.

Some of the people, agencies and businesses that may receive and use your health information are the research sponsor; representatives of the sponsor assisting with the research; investigators at other sites who are assisting with the research; central laboratories, reading centers or analysis centers; the Institutional Review Board; representatives of Wake Forest University Health Sciences and North Carolina Baptist Hospital; representatives from government agencies such as the Food and Drug Administration (FDA) or the Office of Human Research Protections (OHRP), the Department of Health and Human Services (DHHS) and similar agencies in other countries.

Some of these people, agencies and businesses may further disclose your health information. If disclosed by them, your health information may no longer be covered by federal or state privacy regulations. Your health information may be disclosed if required by law. Your health information may be used to create information that does not directly identify you. This information may be used by other researchers. You will not be directly identified in any publication or presentation that may result from this study unless there are photographs or recorded media which are identifiable.

Monitors, auditors, IRB or other regulatory agencies will be granted direct access to the participant's original medical record for verification of clinical trial procedures or data, without violating confidentiality of the participant and to the extent permitted by other applicable laws.

If required by law or court order, we might also have to share your Protected Health Information with a judge, law enforcement officer, government agencies, or others. If your Protected Health Information is shared with any of these groups it may no longer be protected by federal or state privacy rules.

Any Protected Health Information collected from you in this study that is maintained in the

Version: 01/21/20 



research records will be kept for at least six years after the study is finished. At that time any research information not already in your medical record will either be destroyed, or it will be deidentified.

You can tell Michael G. Kelly, M.D. that you want to take away your permission to use and share your Protected Health Information at any time by sending a letter to this address:



However, if you take away permission to use your Protected Health Information you will not be able to be in the study any longer. We will stop collecting any more information about you, but any information we have already collected can still be used for the purposes of the research study.

By signing this form you give us permission to use your Protected Health Information for this study.

If you choose to participate in this study, your medical record at Wake Forest University Baptist Medical Center will indicate that you are enrolled in a clinical trial. Information about the research and any medications or devices you are being given as a participant may also be included in your medical record. This part of the medical record will only be available to people who have authorized access to your medical record. If you are not a patient at this Medical Center, a medical record will be created for you anyway to ensure that this important information is available to doctors in case of an emergency.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this Web site at any time.

Laboratory test results and other medical reports created as a result of your participation in the research study may be entered into the computer systems of Wake Forest University Health Sciences and North Carolina Baptist Hospital. These will be kept secure, with access to this information limited to individuals with proper authority, but who may not be directly involved with this research study.

A North Carolina Baptist Hospital (NCBH) medical record will be created for all study participants. Information about your participation in the study will be placed in the NCBH medical record, along with any routine medical test results that were obtained at NCBH as part of this study.

# WHAT ARE MY RIGHTS AS A RESEARCH STUDY PARTICIPANT?

Taking part in this study is voluntary. You may choose not to take part or you may leave the study at any time. Refusing to participate or leaving the study will not result in any penalty or loss of benefits to which you are entitled. If you decide to stop participating in the study we Version: 01/21/20




encourage you to talk to the investigators or study staff first to learn about any potential health or safety consequences. The investigators also have the right to stop your participation in the study at any time. This could be because it is in your best medical interest, your condition worsened, new information becomes available, you had an unexpected reaction, you failed to follow instructions or procedures, or because the entire study has been stopped.

Version: 01/21/20 